CLINICAL TRIAL: NCT05261750
Title: Safety and Efficacy of Adjuvant Therapy of Autologous Dendritic Cells and Allogenic Dendritic Secretomes for Patients With Advanced Nasopharyngeal Cancer
Brief Title: Autologous Dendritic Cells and Allogenic Dendritic Secretomes for Patients With Advanced Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT/NPC/PSI/2022
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Nasopharyngeal Cancer
Keywords: Dendritic Cells; Dendritic Secretomes
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auto-Dendritic Adjuvant Therapy (Experimental): Patients will be given standard medical therapy (radiotherapy or chemoradiation) and auto-dendritic adjuvant therapy via intramuscular 3 times injection every 1 week.
  Interventions: Biological: Auto-Dendritic Adjuvant Therapy
- Allo-Dendritic-secretome and Auto-Dendritic Adjuvant Therapy (Experimental): Patients will be given standrad medical therapy (radiotherapy or chemoradiation) and allo-dendritic-secretome adjuvant therapy 2 cc 1 times injection, and then followed by auto-dendritic therapy via intramuscular 3 times injection every 1 week.
  Interventions: Biological: Allo-Dendritic-Secretome Adjuvant Therapy

INTERVENTIONS:
Biological: Auto-Dendritic Adjuvant Therapy — Treatment with standard medical therapy (radiotherapy or chemoradiation) and auto-dendritic adjuvant therapy via intramuscular 3 times injection every 1 week.
  Arms: Auto-Dendritic Adjuvant Therapy
Biological: Allo-Dendritic-Secretome Adjuvant Therapy — Treatment with standard medical therapy (radiotherapy or chemoradiation) and allo-dendritic-secretome adjuvant therapy 2 cc 1 times injection, and then followed by auto-dendritic therapy via intramuscular 3 times injection every 1 week.
  Arms: Allo-Dendritic-secretome and Auto-Dendritic Adjuvant Therapy

SUMMARY:
The purpose of this study is to determine the safety and potential of dendritic cells therapy and secretomes therapy for advanced nasopharyngeal cancer.

DETAILED DESCRIPTION:
There are controlled group who receives standard medical theraphy (radiotherapy or chemoradiation), one group who receives standard medical theraphy (radiotherapy or chemoradiation) and Auto-dendritic adjuvant therapy, and other group who receives standard medical theraphy (radiotherapy or chemoradiation) and Allo-dendritic-secretomes adjuvant therapy and continued with auto-dendritic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who tested positive EBV and confirmed suffering advanced nasopharyngeal cancer
* Patients who have partial response or stable disease or progressive disease after performed standard therapy (radiology or chemoradiation) based on RECIST
* Did not take traditional medicine in the last 2 months.
* Patients can understand the nature of the study and willing to sign informed consent
* Patients who received standard medical (radiology or chemoradiation) up to one additional therapy in the last 1 month.

Exclusion Criteria:

* Patients who are pregnant, planning to pregnant, or breastfeeding
* Patients assessed to require chemoradiation during this study
* Patients who get complete score after undergo standard therapy (radiology or chemoradiation) based on the RECIST
* Patients who have autoimun reaction, eczema, allergy or allergy history, and anaphylaxis
* Patients who have creatinin clearance result <40 ml/min, bilirubin serum >1.5x above normal, SGPT-SGOT >5x above normal
* Patients on immunosuppressive medications, such as corticosteroids
* Patients who undergo Major thoracic or abdominal operation
* Patients on high medical risk condition due to uncontrolled infection
* Patients who diagnosed positive of Hepatitis B, Hepatitis C or Human Immunodeificiency virus (HIV)
* Patients who have concurrent congestive heart failure history and other heart disease
* Patients who have health conditions assessed by the doctor in charge cannot be included in this clinical trial
* Patients who refuse or did not participate in part or all of the research process

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Karnofsky Performance Status | Before therapy
  To measure the patient's Quality of Life. Karnofsky Performance Status can be used to determine patient's prognosis and measured changes of patient's ability to do daily activities which ranges from 0-100.
Karnofsky Performance Status | 1 week after therapy
  To measure the patient's Quality of Life. Karnofsky Performance Status can be used to determine patient's prognosis and measured changes of patient's ability to do daily activities which ranges from 0-100.
Karnofsky Performance Status | 1 month after therapy
  To measure the patient's Quality of Life. Karnofsky Performance Status can be used to determine patient's prognosis and measured changes of patient's ability to do daily activities which ranges from 0-100.
Karnofsky Performance Status | 3 months after therapy
  To measure the patient's Quality of Life. Karnofsky Performance Status can be used to determine patient's prognosis and measured changes of patient's ability to do daily activities which ranges from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Rima Haifa, B.Sc, Study Chair — Prodia Stem Cell Indonesia
Locations (1):
- PT Prodia StemCell Indonesia, Jakarta, Indonesia